CLINICAL TRIAL: NCT04365062
Title: Excellent：Clinical Study of Excimer Laser and Drug Coated Balloon Versus Excimer Laser and Plain Balloon Versus Plain Balloon and Drug Coated Balloon to Treat Femoropopliteal In-stent Restenosis
Brief Title: Clinical Study of Excimer Laser and Drug Coated Balloon Versus Excimer Laser and Plain Balloon Versus Plain Balloon and Drug Coated Balloon to Treat Femoropopliteal In-stent Restenosis
Acronym: Excellent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FPA-ISR
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2019-07

CONDITIONS: Atherosclerosis of Artery; In-stent Arterial Restenosis
Keywords: Excimer laser; drug coated balloon; femoropopliteal; In-stent Restenosis
MeSH Terms: interventions — Lasers, Excimer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention: Excimer laser and drug coated balloon (Experimental): Intervention: Excimer laser and drug coated balloon group
  Interventions: Device: Excimer laser and drug coated balloon
- Excimer laser and plain balloon (Active Comparator): Excimer laser and plain balloon group
  Interventions: Device: Excimer laser and plain balloon
- plain balloon and drug coated balloon (Active Comparator): plain balloon and drug coated balloon group
  Interventions: Device: plain balloon and drug coated balloon

INTERVENTIONS:
Device: Excimer laser and drug coated balloon — Excimer laser and drug coated balloon
  Arms: Intervention: Excimer laser and drug coated balloon
Device: Excimer laser and plain balloon — Excimer laser and plain balloon
  Arms: Excimer laser and plain balloon
Device: plain balloon and drug coated balloon — plain balloon and drug coated balloon
  Arms: plain balloon and drug coated balloon

SUMMARY:
This is a randomized study comparing Excimer laser and drug coated balloon Versus Excimer laser and plain balloon versus plain balloon and drug coated balloon to Treat femoropopliteal in-stent restenosis

DETAILED DESCRIPTION:
This is a randomized study comparing Excimer laser and drug coated balloon Versus Excimer laser and plain balloon versus plain balloon and drug coated balloon to Treat femoropopliteal in-stent restenosis

ELIGIBILITY:
Inclusion Criteria:

Provides written informed consent Willing to comply with follow-up evaluations at specified times Has claudication or rest pain due to peripheral arterial In-stent restenosis Disease located within the femoropopliteal artery Patient has a In-stent restenosis lesion(s) with >50% stenosis documented angiographically Patient has symptoms of peripheral arterial disease classified as Rutherford Category 2 or greater.

Exclusion Criteria:

They were excluded if they had one or more of the following: 1. Acute or subacute lower limb ischemia; 2. Severe calcification lesions; 3. Total occlusions lesions more significant than 10 cm or total occlusion lesions with a suspicion of subintimal wire recanalization 4. untreated ipsilateral iliac artery stenosis>70%, or the distal runoff artery <1 root; 5. Previously lower extremity intervention or surgical graft artery bypass; 6. Severe renal insufficiency, creatinine level greater than 2.5 mg/dL; 7. The patient's platelet count is less than 100,000/uL, antiplatelet or anticoagulant contraindications to required medications; 8. Patients with immune system diseases or malignant tumours; 9. ongoing active infection 10. decompensated congestive heart failure or acute coronary syndrome; 11. Unwillingness to return for future follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Primary Patency Rate | 12 months
  Primary patency is defined as no significant reduction of flow detectable by Duplex ultrasound through the index lesion and no further clinically driven target vessel revascularization performed in the interim. Significant reduction of flow is binary restenosis defined as the diameter stenosis >50% with a peak systolic velocity ratio >2.4 as measured by Duplex ultrasound.

SECONDARY OUTCOMES:
Technical success | 1 day
  Technical success is defined as residual stenosis less than 30% by final angiography and/or a flow-limiting dissection.
freedom from clinically-driven TLR | 12 months
  it is defined as freedom from clinically-driven target lesion revascularization
Major Adverse Events | 12 months
  Major adverse events included death, index limb ischemia, index limb amputation, and significant embolic events, which were defined as causing end-organ damage.
Limb Salvage Rate | 12 months
  Limb Salvage is defined as the freedom from secondary major amputation

CONTACTS AND LOCATIONS:
Locations (1):
- Gu Yong Quan, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yongquan G, Lianrui G, Lixing Q, Xuefeng L, Zhu T, Shijun C, Yingfeng W, Jianming G, Jian Z, Zhonggao W. Plaque excision in the management of lower-limb ischemia of atherosclerosis and in-stent restenosis with the SilverHawk atherectomy catheter. Int Angiol. 2013 Aug;32(4):362-7. PMID 23822938